CLINICAL TRIAL: NCT01732276
Title: Phase Ⅱ Study of Gefitinib in Triple-negative,EGFR Positive Metastatic Breast Cancer
Brief Title: The Safety and Effects of Gefitinib in Triple-negative,EGFR Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangmen Central Hospital (Other)
Responsible Party: Principal Investigator, yu gengsheng, vice director of oncology department, Jiangmen Central Hospital, Jiangmen Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120314
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
Keywords: Triple-negative breast cancer; Epidermal growth factor receptor; Gefitinib
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gefitinib (Experimental): gefitinib tablet 250mg/day by mouth until disease progression
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: gefitinib
  Other Names: IRRESA

SUMMARY:
Breast cancer is a heterogeneous disease and can be classified into several distinctive subgroups. Triple-negative breast cancer(TNBC) is defined by lack of estrogen(ER), progesterone(PR) immunoreactivity and lack of human epidermal receptor-2(HER2) overexpression. TNBC comprises around 15% of all breast cancer and is characterized by its aggressive clinical behavior and insensitivity toward available targeted treatment strategies such as endocrine and anti-HER2 therapies.Although TNBC is sensitive to chemotherapy,early relapse with metastatic disease is common and the prognosis is poor. Development Of novel treatment strategies is,therefore,needed and the study of other potential targets in TNBC,like tyrosine kinase receptors,is a topic of interest.

Epidermal Growth Factor Receptor(EGFR) is a transmembrane receptor tyrosine kinase that encoded by cell erythroblastosis virus oncogene B1(C-erbB1) and belongs to the HER/Erythroblastosis virus oncogene B(ErbB) family. By several signal pathways,EGFR regulates cell proliferation, differentiation, apoptosis, invasion,and angiogenesis,and serves as a poor prognostic factor.EGFR is overexpressed in a variety of malignancies including TNBC.Gene expression profiling and immunohistochemical studies have indicated that 40 to 60% of TNBCs exhibit EGFR expression and gene amplification was found in 18% of this subgroup,but EGFR mutation was rare in TNBC.

By far,the role of gefitinib, an EGFR tyrosine kinase inhibitor(TKI),in the metastatic TNBC has not been identified. Most clinical trials about EGFR TKIs in the breast cancer have one or more limitations including:1) the study population had received heavily pretreatment; 2)the enrolled patients included several subgroups of breast cancer; 3)the expression of EGFR was not clear in the enrolled patients.

Here, the investigators launch a prospective clinical trial, and about 50 patients with triple-negative,EGFR positive metastatic breast cancer that have received at least second line therapy will be enrolled. these patients will be treated with gefitinib, the toxicity and effects of gefitinib will be recorded prospectively to evaluate the role of gefitinib in the metastatic TNBC.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* ≥1 measurable or assessable lesion
* Eastern Cooperative Oncology Group(ECOG)performance status of 0-2
* adequate renal,hepatic and hematological function
* a life expectancy of >12 weeks
* histologically proven EGFR positive metastatic TNBC

Exclusion Criteria:

* brain metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
clinical benefit rate | one month
  The primary end point is objective clinical benefit rate defined as objective response or stable disease for≥24wk

SECONDARY OUTCOMES:
progress-free survival（PFS） | every 4 weeks
  Progress-free survival（PFS）is defined as the time from start of treatment to progression or death.

OTHER OUTCOMES:
Toxicity | twice weekly
  Toxicity is assessed twice weekly and adverse effects(AEs) are classified according to the National Cancer Institute Common Toxicity Criteria(NCI-CTC).

CONTACTS AND LOCATIONS:
Overall Officials: gengsheng yu, Principal Investigator — Department of oncology, Jiangmen central hospital, Jiangmen, China